CLINICAL TRIAL: NCT06058065
Title: Value of Xpert® MTB/RIF Ultra in Cases With Suspected Tuberculosis
Brief Title: Sensitivity and Specificity of Xpert MTB/RIF Ultra
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, Lecture of chest diseases, Assiut University
Other Study IDs: Ultra Xpert® MTB/RIF
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To estimate diagnostic accuracy of Xpert Ultra and Xpert MTB/RIF for extrapulmonary tuberculosis and rifampicin resistance in adults suspected to be infected with mycobacterium tuberculosis. In addition, this study will estimate the pattern of rifampicin resistance among TB cases in Assiut population.

DETAILED DESCRIPTION:
Xpert MTB/RIF was introduced recently and added great benefit in management of TB. Xpert MTB/RIF revolutionized the management of Mycobacterium tuberculosis (MTB) infections by providing faster and more accurate MTB diagnosis that detects MTB and rifampicin (RIF) resistance simultaneously. Following World Health Organization (WHO) endorsement in 2010, Xpert MTB/RIF has helped improve TB programs in over 130 countries5.

Building on this success, faster and more accurate detection of MTB from the first point of encounter in the community is critical. Partnered with GeneXpert® Systems, Xpert MTB/RIF Ultra was delivered with the advantages of improved performance and faster time to result (results within 80 minutes). It has higher sensitivity especially in smear-negative TB cases. The processing of the new assay is easy to use and does not need special expertise5. Xpert MTB/RIF Ultra has increased accuracy of Rifampicin results and improved detection of mixed infections. Recently published recommendations by global experts demonstrate the efficiency of using Xpert MTB/RIF Ultra as a frontline test over smear microscopy or line probe assays followed by culture-based methods for drug susceptibility testing. Thus, a single modification of the diagnostic algorithm to detect smear-positive and smear-negative TB patients improves active case management, is more cost-efficient and could potentially reduce the relative rate of transmission. Using Xpert MTB/RIF Ultra has the potential to reduce the number of missed smear-negative TB patients and may lead to a decrease in total costs of patient care due to the detection of MTB in patient specimens and RIF-resistance in a single test. There is great need for further research to assess the diagnostic value of Xpert MTB/RIF Ultra in patients with pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

- Patients presented to Chest Department with suspected pulmonary or extrapulmonary Tuberculosis will be sequentially included

Exclusion Criteria:

* Age: less than 18 years. Patients who received anti tuberculous drugs in the past 6 months. Unstable patients or need for ICU admission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to Assiut University Hospital with suspected Tuberculosis from July 2023 to June 2024 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-11 (Estimated); Primary Completion 2024-11-28 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Xpert MTB/RIF Ultra | Baseline
  By compare with other test

SECONDARY OUTCOMES:
Prevalence of rifampicin resistance among patients with TB active infection presented to Chest Department in Assiut University Hospital | base line
  from results

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed yassen, MD, Study Chair — Assiut University; Abd-Elmalek Abd-Elmalek, MD, Study Chair — Assiut Chest Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kay AW, Ness T, Verkuijl SE, Viney K, Brands A, Masini T, Gonzalez Fernandez L, Eisenhut M, Detjen AK, Mandalakas AM, Steingart KR, Takwoingi Y. Xpert MTB/RIF Ultra assay for tuberculosis disease and rifampicin resistance in children. Cochrane Database Syst Rev. 2022 Sep 6;9(9):CD013359. doi: 10.1002/14651858.CD013359.pub3. PMID 36065889
- [Result] Park M, Kon OM. Use of Xpert MTB/RIF and Xpert Ultra in extrapulmonary tuberculosis. Expert Rev Anti Infect Ther. 2021 Jan;19(1):65-77. doi: 10.1080/14787210.2020.1810565. Epub 2020 Sep 24. PMID 32806986